CLINICAL TRIAL: NCT06528457
Title: A Phase 2, Randomized, Double Blind, Placebo-Controlled Study to Examine the Prophylactic and Treatment Effects of a Single Dose Level of Oral Fenretinide in a Dengue Virus Challenge Model
Brief Title: Study to Examine the Effects of Oral Fenretinide
Acronym: PROTECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Island Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISLA101-P02-CT002
Record Dates: First submitted 2024-07-15; First posted 2024-07-30 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Dengue
Keywords: dengue; Dengue with Warning Signs; Dengue Without Warning Signs
MeSH Terms: conditions — Dengue | interventions — Fenretinide

STUDY DESIGN:
Intervention Model Description: This double-blinded study is designed to examine two potential uses of ISLA101, the first being prophylaxis against infection and the second being treatment of established infection.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental): The first cohort (Cohort A) allows examination of prophylaxis as well as treatment, as ISLA101 will be taken prior to inoculation and for 21 days thereafter. Subjects will be randomized 3:1 (active:control), enrolling in a single group three days prior to inoculation. Following the morning dose on the 4th day of dosing, all subjects will be administered 0.5 mL DENV-1-LVHC (6.5 x 103 PFU/mL).
  Interventions: Drug: ISLA101; Drug: Dengue 1 Live Virus Human Challenge (DENV-1-LVHC)
- Cohort B (Placebo Comparator): The first cohort (Cohort B) allows examination of prophylaxis as well as treatment, as placebo will be taken prior to inoculation and for 21 days thereafter. Subjects will be randomized 3:1 (active:control), enrolling in a single group three days prior to inoculation. Following the morning dose on the 4th day of dosing, all subjects will be administered 0.5 mL DENV-1-LVHC (6.5 x 103 PFU/mL).
  Interventions: Drug: Dengue 1 Live Virus Human Challenge (DENV-1-LVHC); Other: Placebo
- Cohort C (Experimental): The second cohort (Cohort C) is planned to enroll in two groups of five subjects each, using 4:1 randomization (active:control). All subjects will be administered 0.5 mL DENV-1-LVHC (6.5 x 103 PFU/mL) on Day 1. After the inoculation, subjects will be evaluated in the clinic daily through day 18 (eighteen consecutive daily clinic visits). Dosing with ISLA101 will commence on the morning of Day 8 and continue with a total of 28 doses taken twice daily through Day 21.
  Interventions: Drug: ISLA101; Drug: Dengue 1 Live Virus Human Challenge (DENV-1-LVHC)
- Cohort D (Placebo Comparator): The second cohort (Cohort D) is planned to enroll in two groups of five subjects each, using 4:1 randomization (active:control). All subjects will be administered 0.5 mL DENV-1-LVHC (6.5 x 103 PFU/mL) on Day 1. After the inoculation, subjects will be evaluated in the clinic daily through day 18 (eighteen consecutive daily clinic visits). Dosing with placebo will commence on the morning of Day 8 and continue with a total of 28 doses taken twice daily through Day 21.
  Interventions: Drug: Dengue 1 Live Virus Human Challenge (DENV-1-LVHC); Other: Placebo

INTERVENTIONS:
Drug: ISLA101 — ISLA101 is an oral gelatin capsule containing 100 mg of fenretinide (N-[4-Hydroxyphenyl]retinamide, mw 391.56) dissolved in corn oil and polysorbate 80. ISLA101 capsules will be administered orally as one dose of 300 mg/m2 each 12 hours (q12 +/-1 h).
  Other Names: fenretinide
  Arms: Cohort A; Cohort C
Drug: Dengue 1 Live Virus Human Challenge (DENV-1-LVHC) — The DENV-1-LVHC investigational challenge material consists of the dengue-1 virus strain 45AZ5 as a powder, lyophilized for reconstitution. The product is reconstituted with 0.7 mL of water for injection (WFI) and diluted to a concentration of 6.5 x 103 PFU/mL.
Other: Placebo — Placebo capsules will be administered orally as one dose of 300 mg/m2 each 12 hours (q12 +/-1 h).
  Arms: Cohort B; Cohort D

SUMMARY:
This randomized, placebo controlled single center study examines the extent to which 600 mg/m2/day of orally administered ISLA101 (fenretinide), given prophylactically or therapeutically, may reduce or eliminate signs and symptoms of dengue virus (DENV) infection over 29 days following subcutaneous challenge of healthy subjects with 'Dengue 1 Live Virus Human Challenge' (DENV-1-LVHC). Humoral and cellular immune responses, both innate and adaptive, circulating virus, and changes in clinical laboratory measures will also be examined.

DETAILED DESCRIPTION:
Pharmacology studies have identified the potential for fenretinide to inhibit the binding of the DENV nonstructural protein 5 (NS5) to host nuclear importins (IMPs) IMP-α and IMP-β1, thereby impairing infection and replication. This Phase 2 study is to evaluate the effectiveness of fenretinide in an encapsulated oral formulation (ISLA101) against challenge with Dengue 1 Live Virus Human Challenge (DENV-1-LVHC) product, both prophylactically and therapeutically. Oral doses will be taken with a high fat meal to improve absorption, as fenretinide is known to have poor gut permeability attributed to its accumulation in lipophilic cell membranes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects not of childbearing potential who are 18 years to 55 years of age (inclusive) at the time of consent
* Females not of childbearing potential as defined in the following criteria:

  1. History of hysterectomy
  2. Post-menopausal:

  i. Natural post-menopausal females with at least 12 months from natural spontaneous amenorrhea and a serum follicle-stimulating hormone (FSH) concentration ≥ 40 IU/L ii. Post-surgical females must have undergone bilateral oophorectomy at least 6 weeks prior to study
* Male subjects with female partners of childbearing potential must agree to practice abstinence or use a combination of 2 of the following acceptable birth control methods during the study and for at least 90 days after dosing:

  1. Partners with an intrauterine device (IUD) in place for at least 3 months
  2. Barrier method (condom or diaphragm) for at least 14 days prior to screening
  3. Partners using stable hormonal contraceptive for at least 3 months prior to the study
  4. History of vasectomy at least 3 months prior to signing the Informed Consent Form
* Ability and willingness to sign informed consent
* Passing score on comprehension test of at least 75%, with up to 3 attempts
* Available for the study period
* Provide consent for release of medical records from primary care physician, college or university, urgent care or emergency room visit

Exclusion Criteria:

* Known or suspected pregnancy (confirmed via a positive serum human chorionic gonadotropin (hCG) pregnancy test at screening), planned pregnancy during the study period, nursing, or lactation
* Men who intend to father a child or donate sperm during the study period, and for 90 days after dosing with study drug
* Any disorders of coagulation
* Any current malignancy other than non-melanoma skin cancer
* Men who intend to father a child during the study period (approximately 120 days)
* Blood tests confirming infection with human immunodeficiency virus- 1 (HIV-1), hepatitis C, hepatitis B (assessed by HBsAg) virus, or suspicion of active influenza virus infection
* Positive antibodies to dengue virus
* Any history of dengue infection or dengue vaccination (licensed or experimental); or planned dengue vaccination during the study period
* Recent (in the past 4 weeks) travel to any dengue endemic area or travel to a country with risk of Yellow Fever or Japanese encephalitis transmission
* Positive urine screen for cocaine, amphetamines, opiates or methadone
* Currently taking anti-coagulant medication, aspirin or non-steroidal anti-inflammatory drugs (NSAIDs)
* Active diabetes, active peptic ulcer disease (PUD), chronic obstructive pulmonary disease (COPD), coronary artery disease (CAD)
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunomodulation therapy such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Use of drugs listed in §6.6 that inhibit or induce Cytochrome P450 3A4 (CYP 3A4) enzymes within 30 days prior to administration of study drug and for the duration of Subject participation
* Current, or a history of, auto-immune disease other than well controlled Hashimoto's thyroiditis
* History of Guillain-Barré syndrome
* Diagnosis with Bipolar Disorder or Schizophrenia, hospitalization in the past year for a mental health disorder, or any other psychiatric condition, which in the opinion of the investigator prevents the Subject from participating in the study
* Hives, shortness of breath, swelling of the lips or throat, or hospitalization related to a previous vaccination or an allergy to specific medications/animals for which antigens may be in the virus preparations to include: shellfish allergy, fetal bovine serum, L-glutamine, neomycin and streptomycin
* Chronic migraine headaches, defined as more than 15 headache days per month over a 3-month period of which more than 8 are migraines, in the absence of medication over use
* Planning to donate blood in the 1 year following inoculation with dengue
* Recent blood donation within prior 14 days of inoculation
* Receipt of blood products or antibodies within 56 days of inoculation or during the study period
* Planned travel during the study period (~120 days) which would interfere with the ability to complete all study visits
* Any laboratory abnormalities prior to inoculation for the tests specified in the protocol, that are considered by the investigator to be clinically significant except those listed in exclusion criteria #25
* subjects with the following grade 2 or greater lab abnormalities: Creatinine; Liver Function Tests - alanine transaminase (ALT), aspartate aminotransferase (AST); Hemoglobin (females and males); white blood count (WBC) decrease; Platelets decreased; prothrombin time (PT); partial thromboplastin time (PTT); Fibrinogen decrease
* Significant screening physical examination abnormalities at the discretion of the investigator
* Participation (active or follow-up phase) or planned participation in another vaccine, drug, medical device, or medical procedure clinical trial in the 4 weeks prior to this trial or during the trial.
* Recent or scheduled receipt of any vaccine 4 weeks prior to or after virus inoculation
* Beliefs that restrict the administration of blood products or transfusions
* Chronic medical condition that, in the opinion of the investigator, impacts Subject safety
* Physician discretion

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Characterization of DENV viremia following inoculation | over 29 days from inoculation
  Area under the curve of RNAemia by qRT-PCR for Cohort 1
  Time to loss of detection of dengue virus RNAemia for Cohort 2

SECONDARY OUTCOMES:
To further characterize circulating virus in the two interventional groups versus control | over 29 days from inoculation
  Time to positive RNAemia by qRT-PCR
To characterize circulating virus in the two interventional groups versus control | over 29 days from inoculation
  Peak level of RNAemia by qRT-PCR
To characterize circulating virus in the two interventional groups versus control | Over 29 days from inoculation
  Duration of RNAemia by qRT-PCR (Cohort 1)
To characterize circulating virus in the two interventional groups versus control | Over 29 days from inoculation
  Area under the curve of RNAemia by qRT-PCR (Cohort 2)
To characterize circulating virus in the two interventional groups versus control | Over 29 days from inoculation
  Levels of infectious virus in blood by Plaque Assay
To determine the effect of ISLA101 on solicited signs and symptoms of DENV when given prophylactically and through Day 21 post-inoculation, or only as delayed therapy | Over 29 days from inoculation
  The calculated score of solicited signs and symptoms associated with dengue virus infection, including any of the listed events below, will consist of summing the CTCAE grades across all days for all events, where the score will be summarized by number of positive subjects:
  * Fever, nausea, vomiting, fatigue, rash, abdominal pain, eye pain, bone pain, joint pain, muscle pain, headache.
To compare the occurrence of unanticipated signs or symptoms of severe dengue | Over 29 days from inoculation
  The proportion of subjects with any of the following:
  * diffuse abdominal pain or tenderness,
  * persistent vomiting,
  * clinical fluid accumulation (ascites, pleural effusion),
  * mucosal bleeding,
  * lethargy,
  * restlessness,
  * liver enlargement >2 cm,
  * increase in hematocrit concurrent with rapid decrease in platelet count.
  * severe plasma leakage,
  * severe hemorrhage,
  * severe organ impairment.
To compare the need for hospital care between groups | Over 29 days from inoculation
  Proportion of subjects hospitalized for dengue symptoms
To compare the need for hospital care between groups | Over 29 days from inoculation
  Length of hospitalization stay for dengue symptoms
To compare the need for hospital care between groups | Over 29 days from inoculation
  Number of days in the intensive care unit for each hospitalization for dengue symptoms
To evaluate changes from baseline in platelet among the three groups | Over 29 days from inoculation
  Number of participants with abnormal platelet counts, observed over 29 days from inoculation, will be summarized overall, by group, by duration and by toxicity grade for each group compared with control. A summary of subjects with shifts from baseline (relative to normal range) in laboratory test results will be provided.
To describe the Cmax of ISLA101 at the tested dose, route, and duration | from first to next to last dose of ISLA101 (Day 24) for Cohort 1
  Concentration-time plots of first and NEXT-TO-LAST dose of ISLA101
To describe the Tmax of ISLA101 at the tested dose, route, and duration | from first to next to last dose of ISLA101 (Day 24) for Cohort 1
  Concentration-time plots of first and NEXT-TO-LAST dose of ISLA101
To describe the Cmax of ISLA101 at the tested dose, route, and duration | from first to next to last dose of ISLA101 (Day 21) for Cohort 2
  Concentration-time plots of first and NEXT-TO-LAST dose of ISLA101
To describe the Tmax of ISLA101 at the tested dose, route, and duration | from first to next to last dose of ISLA101 (Day 21) for Cohort 2
  Concentration-time plots of first and NEXT-TO-LAST dose of ISLA101

CONTACTS AND LOCATIONS:
Overall Officials: Bert Slade, MD, Study Director — CCRS
Locations (1):
- SUNY Upstate Medical University, East Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No